CLINICAL TRIAL: NCT02140580
Title: Multicentre Randomised Controlled Trial of Minimally-invasive Surfactant Therapy in Preterm Infants 25-28 Weeks Gestation on Continuous Positive Airways Pressure
Brief Title: OPTIMIST-A Trial: Minimally-invasive Surfactant Therapy in Preterm Infants 25-28 Weeks Gestation on CPAP
Acronym: OPTIMIST-A
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Menzies Institute for Medical Research (Other)
Collaborators: Royal Hobart Hospital (Other Government); Royal Women's Hospital, Melbourne, Australia (Unknown); Endeavor Health (Other); Monash Medical Centre (Other); Mercy Hospital for Women, Australia (Other); Auckland City Hospital (Other Government); Middlemore Hospital, New Zealand (Other); Zekai Tahir Burak Women's Health Research and Education Hospital (Other); Kapiolani Medical Center For Women & Children (Other); The Cooper Health System (Other); Yale University (Other); West Virginia University Hospital (Unknown); Uludag University (Other); Ziv Medical Center (Other); Bnai Zion Medical Center (Other Government); University Medical Centre Ljubljana (Other); Dunedin Hospital (Other); Kanuni Sultan Suleyman Training and Research Hospital (Other); University Medical Center Groningen (Other); University of Southern California (Other)
Responsible Party: Principal Investigator, Professor Peter Dargaville, Consultant Neonatologist, Paediatric and Neonatal Intensive Care Unit, Royal Hobart Hospital, Menzies Institute for Medical Research
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 4.3, 6th June 2013
Record Dates: First submitted 2014-05-13; First posted 2014-05-16 (Estimated); Last update posted 2020-05-01 (Actual); Status verified 2020-04

CONDITIONS: Bronchopulmonary Dysplasia
Keywords: Minimally-invasive surfactant therapy
MeSH Terms: conditions — Bronchopulmonary Dysplasia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Minimally invasive surfactant therapy (Active Comparator): Minimally invasive surfactant therapy - delivery of exogenous surfactant to the lung via brief catheterisation of the trachea with an instillation catheter in a preterm infant who is being supported with continuous positive airway pressure (CPAP) via nasal prongs or mask. Poractant alfa (Curosurf) at a dosage of 200 mg/kg will be administered over 15 - 30 seconds. Total duration of the procedure will be less than 5 minutes, followed by reinstitution of CPAP.
  Interventions: Device: Minimally invasive surfactant therapy
- Continuation on CPAP (Sham Comparator): Standard control treatment. After randomisation, infants will receive a sham treatment from a treatment team not engaged in clinical care. This will not involve removal of prongs or discontinuation of CPAP but will require setting up intubation equipment, screening the baby, testing suction unit, repositioning of the baby and changing the baby's monitoring. CPAP will thereafter continue.
  Interventions: Other: Continuation on CPAP

INTERVENTIONS:
Device: Minimally invasive surfactant therapy — Active Comparator
  Other Names: 16G Angiocath, Product No. 382259, BD, Sandy, UT, USA
  Arms: Minimally invasive surfactant therapy
Other: Continuation on CPAP — Sham Comparator
  Other Names: Standard care - continuation of CPAP
  Arms: Continuation on CPAP

SUMMARY:
Trial question: Does administration of exogenous surfactant using a minimally-invasive technique improve outcome in preterm infants 25-28 weeks gestation treated with continuous positive airway pressure (CPAP)? Trial hypothesis: That early surfactant administration via a minimally-invasive technique to preterm infants on CPAP will result in a lesser duration of mechanical respiratory support, and a higher incidence of survival without bronchopulmonary dysplasia. Trial design: Multicentre, randomised, masked, controlled trial in inborn preterm infants 25-28 weeks gestation, aged less than 6 hours, requiring CPAP because of respiratory distress, with an FiO2 of >=0.3 and CPAP pressure 5-8. Infants randomised to surfactant treatment receive 200 mg/kg of poractant alfa (Curosurf) administered under direct laryngoscopy using a surfactant instillation catheter, followed by reinstitution of CPAP. Controls continue on CPAP. The intervention is masked from the clinical team. Care thereafter is as per usual in both groups, other than the requirement to adhere to intubation criteria. The primary outcome is incidence of death or BPD. Secondary outcomes include incidence of death, major neonatal morbidities (BPD, intraventricular haemorrhage, periventricular leukomalacia, retinopathy of prematurity, necrotising enterocolitis), pneumothorax and patent ductus arteriosus; need for intubation and surfactant therapy; durations of mechanical respiratory support, intubation, CPAP, intubation and CPAP, high flow nasal cannula (HFNC), oxygen therapy, intensive care stay and hospitalisation; hospitalisation cost; applicability and safety of the MIST procedure; and outcome at 2 years. The sample size is 303/group, allowing detection of a 33% difference in the primary outcome with 90% power. The trial commenced at Royal Hobart Hospital December 2011 and Royal Women's Hospital during 2012, and will ultimately be conducted over 5 years in multiple centres internationally.

DETAILED DESCRIPTION:
1. OPTIMIST-A TRIAL SUMMARY RESEARCH QUESTION Does administration of exogenous surfactant using a minimally-invasive technique improve outcome in preterm infants 25-28 weeks gestation treated with continuous positive airway pressure (CPAP)?

BACKGROUND Nasal CPAP is often very effective in preterm infants as the initial means of respiratory support, but a sub-group of infants, most with features of respiratory distress syndrome, fail on CPAP and require intubation and ventilation in the first 72 hours. When compared to those in whom CPAP is successful, infants failing CPAP have a substantially longer duration of respiratory support, and a higher risk of adverse outcomes. Decreasing the risk of CPAP failure would thus seem advantageous, and may be achievable with minimally invasive surfactant therapy (MIST), in which surfactant is administered to a spontaneously breathing infant who then remains on CPAP. A technique of MIST (the "Hobart method") using a semi-rigid surfactant instillation catheter has been shown to be feasible in preterm infants on CPAP, and appears to have the potential to alter respiratory course and outcome. This method of MIST now requires evaluation in randomised controlled trials.

RESEARCH DESIGN Multicentre, randomised, masked, controlled trial.

RECRUITMENT Entry criteria Inborn preterm infants 25-28 weeks gestation, aged less than 6 hours, who were not intubated at birth but require CPAP or NIPPV because of respiratory distress, with a CPAP pressure of 5-8 cm H2O and FiO2 ≥0.30.

Exclusion criteria Infants will be excluded if in imminent need of intubation, or if there is a congenital anomaly or alternative cause for respiratory distress.

RANDOMISATION With parental consent, eligible infants will be randomly allocated using a web-based randomisation server, with stratification by study centre, to receive exogenous surfactant via the Hobart MIST technique, or to continue on CPAP.

INTERVENTION Infants randomised to surfactant treatment will receive a dose of poractant alfa (Curosurf) administered under direct laryngoscopy using a surfactant instillation catheter, at a dosage of 200 mg/kg. CPAP will thereafter be reinstituted. Controls will continue on CPAP. The intervention will be masked from the clinical team.

POST-INTERVENTION MANAGEMENT Other than the requirement to adhere to intubation criteria in the first week, and in some cases perform a room air trial at 36 weeks corrected gestation, management after intervention will be at the discretion of the clinical team. Titration of CPAP pressure is encouraged, with a permitted maximum of 8 cm H2O. Nasal IPPV (bi-level CPAP) is allowable. Early caffeine therapy is expected.

Criteria for intubation: Enrolled infants on CPAP will be intubated if FiO2 ≥0.45, or if there is unremitting apnoea or persistent acidosis. These criteria apply during the first week of life, and to the first episode of intubation only.

FOLLOWUP: At 2 years corrected age, parents of each infant will complete a brief health assessment and a validated child development assessment (PARCA-R, Dev Med Child Neurol 2004;46:389-97) administered as a web-based questionnaire located on a secure server. The infant-specific link to the questionnaire, and reminders where necessary, will be sent electronically to the parents by research personnel at each Site, thus maintaining confidentiality. No identifying details will be revealed in the completion of the questionnaire.

OUTCOMES Primary outcome: Incidence of composite outcome of death or physiological bronchopulmonary dysplasia (BPD).

Secondary outcomes: Incidence of death, major neonatal morbidities (BPD, intraventricular haemorrhage, periventricular leukomalacia, retinopathy of prematurity, necrotising enterocolitis), pneumothorax and patent ductus arteriosus; need for intubation and surfactant therapy; durations of mechanical respiratory support, intubation, CPAP, intubation and CPAP, high flow nasal cannula (HFNC), oxygen therapy, intensive care stay and hospitalisation; hospitalisation cost; applicability and safety of the MIST procedure; and outcome at 2 years.

SAMPLE SIZE 606 infants (303 per group), giving 90% power to detect a 33% reduction in death or BPD from the anticipated rate of 38% in the control arm, α = 0.05.

TRIAL PLAN The OPTIMIST trials will commence at RHH Hobart and RWH Melbourne during 2011. All Australasian neonatal units, and selected international centres including those in the Vermont- Oxford Network, will be invited to join the trials. A full complement of participating centres is expected by early 2014. Recruitment will thereafter proceed at full rate until completion, which is estimated to take up to 4 years.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age 25-28 completed weeks
* Requiring CPAP or non-invasive positive pressure ventilation with signs of early respiratory distress.
* CPAP pressure of 5-8 cm H2O and FiO2 >=0.30.
* Less than 6 hours of age.
* Agreement of the Treating Physician in charge of the infant's care.
* Signed parental consent.

Exclusion Criteria:

* Previously intubated, or in imminent need of intubation
* Congenital anomaly or condition that might adversely affect breathing.
* Identifiable alternative cause for respiratory distress (e.g. congenital pneumonia or pulmonary hypoplasia).
* Lack of availability of an OPTIMIST treatment team.

Ages: 1 Minute to 6 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 486 (Actual)
Dates: Start 2011-12; Primary Completion 2020-05 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Death or physiological bronchopulmonary dysplasia | 36 weeks post menstrual age
  Composite outcome of death by 36 weeks or physiological bronchopulmonary dysplasia (BPD). Physiological BPD is assessed at 36 weeks post-menstrual age, and is defined as either need for respiratory support (intubation / CPAP / high flow nasal cannula > 2 L/min) or need for FiO2 >=0.3 or failure of a room air trial conducted at 36 weeks post-menstrual age. This will be assessed by the research nurse at each centre.

SECONDARY OUTCOMES:
Mortality | 36 weeks post menstrual age
Major morbidity | 36 weeks post menstrual age
  Major morbidity, defined as one or more of BPD, grade III or IV intraventricular haemorrhage, periventricular leukomalacia or retinopathy of prematurity > stage 2, occurring at any time up to 36 weeks post menstrual age. Screening for intraventricular haemorrhage, periventricular leukomalacia and retinopathy of prematurity will be performed as routine care, and the results taken from the medical record.
Pneumothorax | 36 weeks post menstrual age
  Pneumothorax at any time up to 36 weeks post menstrual age, as documented in medical record.
Duration of respiratory support | During first hospitalisation (average assessment period 14 weeks)
  Duration of respiratory support, defined as cumulative hours of all episodes of intubation, nasal CPAP and high flow nasal cannula oxygen (flow rate >= 2 litres/min). This information will be derived from medical record or unit database.
Bronchopulmonary dysplasia | 36 weeks post menstrual age
  Bronchopulmonary dysplasia (BPD) will be assessed both clinically (need for mechanical respiratory support and/or an oxygen requirement at 36 weeks corrected gestation), and by a physiological definition. Physiological BPD is assessed at 36 weeks post-menstrual age, and is defined as either need for respiratory support (intubation / CPAP / high flow nasal cannula > 2 L/min) or need for FiO2 >=0.3 or failure of a room air trial conducted at 36 weeks post-menstrual age. This will be assessed by the research nurse at each centre.
Duration of bradycardia and hypoxaemia during intervention | During intervention
  Heart rate and oxygen saturation will be monitored continuously during the intervention. The severity and duration of bradycardia and hypoxia will thus be documented during delivery of exogenous surfactant via brief tracheal catheterisation.
Discomfort during intervention | During intervention
  The incidence of apparent discomfort, as judged by the nurse assisting in the surfactant delivery procedure, will be ascertained in the group randomised to receive surfactant via brief tracheal catheterisation.

OTHER OUTCOMES:
Hospitalisation cost | First hospitalisation (average assessment period 14 weeks)
  The mean of patient billings and mean cost of hospitalisation per patient will be determined, and compared between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Peter A Dargaville, MD, Principal Investigator — Menzies Institute of Medical Research, University of Tasmania
Locations (16):
- United States (5):
  - Yale-New Haven Children's Hospital, New Haven, Connecticut
  - Kapi'olani Medical Center for Women and Children, Honolulu, Hawaii
  - NorthShore Health University HealthSystem Evanston Hospital, Evanston, Illinois
  - Cooper University Hospital, Camden, New Jersey
  - West Virginia University Hospital, Morgantown, West Virginia
- Australia (4):
  - Royal Hobart Hospital, Hobart, Tasmania
  - Royal Womens Hospital, Melbourne, Victoria
  - Mercy Hospital for Women, Melbourne, Victoria
  - Monash Medical Centre, Melbourne, Victoria
- Israel (2):
  - Bnai Zion Medical Center, Haifa
  - Ziv Medical Center, Safed
- New Zealand (2):
  - Auckland City Hospital, Auckland
  - Middlemore Hospital, Auckland
- University Medical Center, Ljubljana, Zaloska, Ljubljana, Slovenia
- Turkey (Türkiye) (2):
  - Uludag University Hospital, Görükle, Bursa
  - Zekai Tahir Burak Hospital, Ankara

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dargaville PA, Aiyappan A, De Paoli AG, Kuschel CA, Kamlin CO, Carlin JB, Davis PG. Minimally-invasive surfactant therapy in preterm infants on continuous positive airway pressure. Arch Dis Child Fetal Neonatal Ed. 2013 Mar;98(2):F122-6. doi: 10.1136/archdischild-2011-301314. Epub 2012 Jun 9. PMID 22684154
- [Background] Dargaville PA, Aiyappan A, Cornelius A, Williams C, De Paoli AG. Preliminary evaluation of a new technique of minimally invasive surfactant therapy. Arch Dis Child Fetal Neonatal Ed. 2011 Jul;96(4):F243-8. doi: 10.1136/adc.2010.192518. Epub 2010 Oct 21. PMID 20971722
- [Background] Dargaville PA. Innovation in surfactant therapy I: surfactant lavage and surfactant administration by fluid bolus using minimally invasive techniques. Neonatology. 2012;101(4):326-36. doi: 10.1159/000337346. Epub 2012 Jun 1. PMID 22940622
- [Derived] Dargaville PA. CPAP, Surfactant, or Both for the Preterm Infant: Resolving the Dilemma. JAMA Pediatr. 2015 Aug;169(8):715-7. doi: 10.1001/jamapediatrics.2015.0909. No abstract available. PMID 26053233
- [Derived] Dargaville PA, Kamlin CO, De Paoli AG, Carlin JB, Orsini F, Soll RF, Davis PG. The OPTIMIST-A trial: evaluation of minimally-invasive surfactant therapy in preterm infants 25-28 weeks gestation. BMC Pediatr. 2014 Aug 27;14:213. doi: 10.1186/1471-2431-14-213. PMID 25164872